CLINICAL TRIAL: NCT06550518
Title: Real-life Second-line Epirubicin-Paclitaxel Regimen as Treatment of Relapsed Small-Cell Lung Cancer : EpiTax Study
Acronym: EPITAX
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC21.0086 - EPITAX
Record Dates: First submitted 2021-06-18; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Advanced Small Cell Lung Carcinoma
Keywords: Small-cell Lung Cancer; Epirubicin; Paclitaxel; Cerebral Efficacy; Real-life
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Initial chemosensitivity is known concerning SCLC but relapse is almost systematic, especially at a metastatic stage. Brain metastasis are identified around 40 to 50% during the evolution of the disease. Concerning the efficacy of epirubicin combined with paclitaxel from the second-line treatment, data is lacking more particularly about specific response on brain metastasis.

In this retrospective multicentric observational study in real life conditions, we try to evaluate systemic and specific cerebral efficacy and safety of a regimen combining epirubicin and paclitaxel in patients treated between 2010 and 2020 for a small cell lung carcinoma from the second-line treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥18 years)
* Histologically or cytologically SCLC diagnosis
* Treated with epirubicin-paclitaxel doublet between January 2010 and December 2020

Exclusion Criteria:

* Opposition to participate registered
* Patients under legal protection
* Patients afflicted by another subtype of lung carcinomas
* SCLC not treated with the epirubicin-paclitaxel doublet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (age ≥18 years) with histologically or cytologically SCLC diagnosis was confirmed who received at least one cycle with a epirubicin-paclitaxel doublet treated between January 2010 and December 2020 in one of the three centers (Brest University Hospital Center, Quimper Hospital Center and Landerneau Hospital Center)
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2021-12-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | through study completion, an average of 1 year
  Time from epirubicin-paclitaxel regimen initiation to disease progression (according to Response Evaluation Criteria In Solid Tumors v1.1) or death from any cause

SECONDARY OUTCOMES:
Overall survival | 1 year
  Time from epirubicin-paclitaxel regimen initiation to death from any cause
Objective response rate | 1 year
  Complete response or partial response (according to Response Evaluation Criteria In Solid Tumors v1.1)
Disease control rate | 1 year
  Objective response rate and stable disease (according to Response Evaluation Criteria In Solid Tumors v1.1)
Intracranial control rate | 1 year
  Objective response rate and stable disease (according to Response Evaluation Criteria In Solid Tumors v1.1)
Toxicities | 1 year
  According to Common Toxicity Criteria for Adverse Events version 5.0.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHRU de Brest, Brest
  - Hôpital de Landerneau, Landerneau
  - CHIC, Quimper

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three month and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.